CLINICAL TRIAL: NCT03085082
Title: Study of the Relationship Between Blood Groups,RH and Skeletal Malocclusion in a Group of Egyptian Population: a Cross Sectional Study
Brief Title: Study of the Relationship Between Blood Groups,RH and Skeletal Malocclusion : a Cross Sectional Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noor Elsebai Mohamed, Master student of the orthodontic program Cairo university, Cairo University
Other Study IDs: skeletal_malocclusion_ABO
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Class II Malocclusion; Class III Malocclusion
MeSH Terms: conditions — Overbite; Malocclusion, Angle Class III | interventions — Blood Grouping and Crossmatching

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- skeletal class II subjects: patients with wits appraisal more than 3 mm measured on a cephalometric x ray obtained during diagnosis
  Interventions: Diagnostic Test: blood type test
- skeletal class III subjects: patients with wits appraisal less than -3 mm measured on a cephalometric x ray obtained during diagnosis
  Interventions: Diagnostic Test: blood type test
- skeletal class I patients: patients with Wits appraisal between -3 and +3 that is measured from a cephalometric x ray obtained during diagnosis of arch length discrepancy. this group will serve as control and obtained after recruitment of the other 2 groups in 1 to 1 fashion
  Interventions: Diagnostic Test: blood type test

INTERVENTIONS:
Diagnostic Test: blood type test — a blood sample will be withdrawn from the subjects tested by anti A anti B and anti D antigens to detect the individuals blood group and RH. then statistical analysis to detect presence of a relationship between skeletal types of malocclusion and ABO blood groups
  Other Names: ABO and RH test; blood typing

SUMMARY:
the study is searching if there is a relationship between the blood groups and RH and the skeletal malocclusion using the skeletal class I as a control group

DETAILED DESCRIPTION:
The study will be conducted on the patients seeking medical care in the orthodontic department Cairo University, for six months all patients with class II and class III malocclusion will be recruited based on Wits appraisal measured from the cephalometric X-ray taken routinely during orthodontic examination. Then a group of class I arch length discrepancy patients will be used as control. A blood sample will be withdrawn and taken to the Cairo university laboratory to analyze the blood group and RH .a statistical analysis will be performed to detect a relationship between skeletal malocclusion and the blood groups as compared to the control

ELIGIBILITY:
Inclusion Criteria:

skeletal class I,II and III patients non syndromic patients above the age of 18 no previous surgical intervention for correction of skeletal malocclusion

Exclusion Criteria:

* syndromic patients
* cleft patients
* patients with previous surgery to correct skeletal malocclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients with skeletal malovclusion seeking medical care in the orthodontic department of cairo university for six months
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
relationship between blood group and skeletal malocclusion | the recruitment will be for six months
  If skeletal malocclusion subjects were found to have a high percentage of a certain blood type or RH when compared to the control group it will be reported that there is a relationship between blood group and skeletal malocclusion. If percentages of blood groups are approximately the same in the malocclusion subjects and the control then the investigator will report that there is no relationship between blood groups and skeletal malocclusion

CONTACTS AND LOCATIONS:
Overall Officials: Amgad qaddah, professor, Study Director — head of department of orthodontics cairo university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flannery, P. M. (1969). Loyola eCommons The Abo Human Blood Groups and Skeletal Class IIi Malocclusions.
- [Background] Schnibben, C. L. (1968). Loyola eCommons A Study of the Relationships of the ABO Human Blood Groups , the Rh Factor and Hereditary Malocclusions of the Skeletal Type , Class II , Division 1.
- [Background] Gheisari R, Ghoreishian M, Movahedian B, Roozbehi A. The association between blood groups and maxillofacial deformities. Indian J Plast Surg. 2008 Jul;41(2):138-40. doi: 10.4103/0970-0358.44921. PMID 19753252
- [Background] Science, D. (2015). International Journal of Pharma and Bio Sciences ISSN CRANIOFACIAL MORPHOLOGY WITH GENETIC INFLUENCE OF ABO BLOOD, 6(4), 412±418.